CLINICAL TRIAL: NCT06174636
Title: Lung Overdistension and Abdominal Pressure Rise: an EIT Based Pilot Study
Brief Title: Lung Overdistension and Abdominal Pressure Rise
Acronym: LOVE BEER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Paolo Persona, Medical Doctor, Principal Investigator, University of Padova
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AOP2978
Record Dates: First submitted 2023-07-09; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Respiratory Failure; Respiratory Distress Syndrome, Adult
Keywords: Abdominal pressure; Overdistension
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Abdominal Pressure Rise (Experimental): Application of an abdominal weight and record of respiratory mechanics data, intra-abdominal pressure variation, Electrical Impedance Tomography data
  Interventions: Procedure: Application of abdominal weight

INTERVENTIONS:
Procedure: Application of abdominal weight — Application of variable weight on the abdomen to reach a 5 mmHg increase in IAP
  Other Names: Intra abdominal pressure rise

SUMMARY:
The goal of this pilot interventional no-profit study is to evaluate airway pressure, esophageal pressure and variations in lung volume distribution with EIT in mechanically ventilated patients admitted to our UTI with respiratory failure after the application of an abdominal weight and resulting increase of intra-abdominal pressure.

ELIGIBILITY:
Inclusion Criteria:

* Invasive mechanical ventilation in acute respiratory failure (PaO2/FiO2 <300 mmHg)
* Need of PEEP trial
* Need of urinary catheter (used to measure IAP)

Exclusion Criteria:

* Contraindication to EIT use
* Pacemaker or other metal device in thoracic region
* Contraindication to abdominal weight placement
* Surgical or traumatic incision on the abdomen
* Severe abdominal hypertension
* Esophageal diseases that counterindicate naso-gastric tube placement
* Severe hemodynamic instability (norepinephrine > 0.1 mcg/kg/min; dobutamine or dopamine > 5 mcg/kg/min; epinephrine every dosage)
* Severe obesity (BMI > 35 kg/m2)
* Need of > 7 kg weight to reach 5 mmHg IAP increase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Variation of lung volume distribution | through study completion, an average of 1 year
  TID %
Variation of airway pressure | through study completion, an average of 1 year
  cmH2O
Variation of esophageal pressure | through study completion, an average of 1 year
  cmH2O

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Università di Padova, Padua, Italy

REFERENCES:
- [Derived] Pacchiarini G, Pettenuzzo T, Zarantonello F, Sella N, Lumetti G, Boscolo A, De Cassai A, Cammarota G, Persona P, Navalesi P; LOVE BEER Study Group. The "mechanical paradox" unveiled: a physiological study. Crit Care. 2025 May 16;29(1):194. doi: 10.1186/s13054-025-05385-9. PMID 40380228